CLINICAL TRIAL: NCT05381675
Title: Short Term Outcomes of Tele-Rehabilitation in Patients With Post-Covid Syndrome
Brief Title: Short Term Results of Tele-Rehabilitation
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Harran University (Other)
Responsible Party: Principal Investigator, Zeynal Yasacı, Research Assistant, Harran University
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: İntervention
Record Dates: First submitted 2022-05-15; First posted 2022-05-19 (Actual); Last update posted 2023-08-29 (Actual); Status verified 2023-08

CONDITIONS: COVID-19; Dyspnea
Keywords: Tele-rehabilitation; COVID-19
MeSH Terms: conditions — COVID-19; Dyspnea

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention (Experimental): Participants will receive a supervised tele-rehabilitation program 2 days a week for 6 weeks.
  Interventions: Other: Tele-rehabillitation
- Control (Other): Participants will receive the same rehabilitation program as prescribed.
  Interventions: Other: Prescribed Exercise Program

INTERVENTIONS:
Other: Tele-rehabillitation — Tele-rehabilitation program will be performed by physiotherapist two times a week for six consecutive weeks. Program including the following exercises:
  Breathing exercises Aerobic exercises Flexibility Strengthening exercises
  Arms: Intervention
Other: Prescribed Exercise Program — The prescribed exercise program will be performed two times a week for six consecutive weeks. Program including the following exercises:
  Breathing exercises Aerobic exercises Flexibility Strengthening exercises
  Arms: Control

SUMMARY:
Most people who have coronavirus disease (COVID-19) recover completely without any sequelae. However, some patients continue to experience symptoms of COVID-19 even though their tests turn negative. This clinical spectrum that occurs after acute infection is called the post-COVID syndrome (PCS). Dyspnea, pain, decreased exercise capacity, limitations in activities of daily living, poor sleep quality, anxiety and depression are common symptoms in PCS. The aim of our study is to examine the effect of tele-rehabilitation-based exercise program on dyspnea, pain, functional capacity, sleep quality, anxiety and depression in individuals with PCS.

ELIGIBILITY:
Inclusion Criteria:

* Being between the ages of 18-75,
* Being in stable medical condition, conscious and cooperative,
* Having had COVID and continuing symptoms
* Volunteering to participate in the study,
* Own a device that can be connected online independently or with support from family members.

Exclusion Criteria:

SpO2 < 92%,

* Hypotension (Systolic Blood Pressure < 90 mmHg or Diastolic Blood Pressure < 60mmHg)
* Having chronic respiratory disease (COPD, Asthma, etc.)
* Having a stroke or neurodegenerative disease.
* Not being willing to participate in the study

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 60 (Actual)
Dates: Start 2022-05-20 (Actual); Primary Completion 2023-05-20 (Actual); Study Completion 2023-08-01 (Actual)

PRIMARY OUTCOMES:
Change from the baseline to the 6th week in mMRC (Modified Medical Research Council) Dyspnoea Scale | Baseline and 6th week
  The mMRC Dyspnoea Scale is used to assess the degree of baseline functional disability due to dyspnoea

SECONDARY OUTCOMES:
Change from the baseline to the 6th week in NPRS | Baseline and 6th week
  The Numerical Rating Scale (NPRS-11) is an 11-point scale for self-report of pain. It is the most commonly used unidimensional pain scale. The respondent selects a whole number (integers 0-10) that best reflects the intensity (or other quality if requested of his/her pain.
Change from the baseline to the 6th week in the 5 times sit to stand test (5XSST) | Baseline and 6th week
  The 5XSST scoring is based on the amount of time (to the nearest decimal in seconds) a patient is able to transfer from a seated to a standing position and back to sitting five times. The equipment need in performing 5XSST test includes: Stopwatch and standard height chair with straight back.
Change from the baseline to the 6th week in the Hospital Anxiety and Depression Scale | Baseline and 6th week
  The Hospital Anxiety and Depression Scale (HADS) was devised to measure anxiety and depression in a general medical population of patients. The questionnaire comprises seven questions for anxiety and seven questions for depression, and takes 2-5min to complete. Although the anxiety and depression questions are interspersed within the questionnaire, it is vital that these are scored separately.
Change from the baseline to the 6th week in the The Pittsburgh Sleep Quality Index | Baseline and 6th week
  The Pittsburgh Sleep Quality Index (PSQI) is a measure of self-reported sleep quality and sleep disturbance. Scoring Using a four-point, Likert-type scale, respondents indicate how frequently they exhibit certain sleep behaviors (0 = "few," 1 = "some- times," 2 = "often," and 3 = "almost always"). The PSQI takes about 10 minutes to complete and it doesn't involve any procedures or interventions.

CONTACTS AND LOCATIONS:
Locations (1):
- İstanbul University-Cerrahpasa, Istanbul, Turkey (Türkiye)

REFERENCES:
- [Derived] Yasaci Z, Mustafaoglu R, Ozgur O, Kuveloglu B, Esen Y, Ozmen O, Yalcinkaya EY. Virtual recovery: efficacy of telerehabilitation on dyspnea, pain, and functional capacity in post-COVID-19 syndrome. Ir J Med Sci. 2025 Apr;194(2):631-640. doi: 10.1007/s11845-025-03899-3. Epub 2025 Feb 8. PMID 39920519